CLINICAL TRIAL: NCT00089128
Title: Phase II Study Of Gemcitabine And CPT-11 (Irinotecan) In Locally Advanced Or Metastatic Bladder Cancer
Brief Title: Gemcitabine and Irinotecan in Treating Patients With Locally Advanced or Metastatic Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000378047; MUSC-100615; PHARMACIA-440EONCO020298; MUSC-HR-10212
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; recurrent bladder cancer; stage III bladder cancer; stage IV bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine and Irnotecan (Experimental)
  Interventions: Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and irinotecan, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with irinotecan works in treating patients with locally advanced or metastatic bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine response in patients with locally advanced or metastatic transitional cell carcinoma of the bladder treated with gemcitabine and irinotecan.

Secondary

* Determine the duration of response in patients treated with this regimen.
* Determine the tolerance to and toxicity of this regimen in these patients.
* Determine the median and progression-free survival of patients treated with this regimen.

OUTLINE: Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with responding disease receive 2 additional courses beyond best response.

Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the bladder

  * Locally advanced or metastatic disease
* Unidimensionally measurable disease by physical exam or imaging study

  * The following are not considered measurable disease:

    * Bone only disease
    * Pleural or peritoneal effusions
    * CNS lesions
    * Irradiated lesions unless disease progression was documented after radiotherapy
* Not amenable to surgery

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 2.0 mg/dL

Renal

* Creatinine ≤ 2.0 mg/dL

Gastrointestinal

* No active inflammatory bowel disease
* No significant bowel obstruction
* No chronic diarrhea

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active malignancy except nonmelanoma skin cancer
* No mental incapacitation or psychiatric illness that would preclude giving informed consent
* No other severe disease that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* No more than 1 prior platinum-based chemotherapy regimen
* At least 4 weeks since prior chemotherapy
* No prior irinotecan or gemcitabine
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormones except steroids for adrenal failure, hormones for non-disease-related conditions (e.g., insulin for diabetes), and intermittent dexamethasone as an antiemetic

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent palliative radiotherapy

Surgery

* Not specified

Other

* No concurrent participation in another clinical trial

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2001-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uzair B. Chaudhary, MD, Study Chair — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine and Irnotecan: On day 1 and day 8 of each 21 day cycle:
  gemcitabine hydrochloride 1,000 mg/m2 IV over 30 minutes
  irinotecan hydrochloride 100mg/m2 IV over 90 minutes
Period: Overall Study
Arm/Group | Gemcitabine and Irnotecan
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine and Irnotecan
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Response Proportion
Time Frame: From registration until time of complete response or partial response
Population: Data for this endpoint was not collected
Arm/Group | Gemcitabine and Irnotecan
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response
Time Frame: From registration until disease progression among patients who had at least a partial response.
Population: Data for this endpoint was not collected
Arm/Group | Gemcitabine and Irnotecan
Number analyzed (Participants) | 0

3. Secondary Outcome: Frequency of Adverse Events as Assessed by NCI CTC Version 2.0
Time Frame: From the day of first dose until the end of study, an average of 6 months
Population: data for this endpoint was not collected
Arm/Group | Gemcitabine and Irnotecan
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Time Frame: Time between registration and disease progression or death, whichever comes first.
Population: data for this endpoint was not collected
Arm/Group | Gemcitabine and Irnotecan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: from start of treatment until end of study, an average of 6 months
Description: The data for this endpoint was not collected
Arm/Group | Gemcitabine and Irnotecan
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes